CLINICAL TRIAL: NCT05420116
Title: Pilot Study of the " Cerdanya on Fitness" Program to Promote the Physical Exercise, Healthy Nutritional Habits and Psycho-emotional Well-being of Obese People in Cerdanya. Pilot Study of the "Cerdanya on Fitness" Program to Promote Physical Exercise, Healthy Nutritional Habits and Psychoemotional Well-being of People With Obesity in Cerdanya.
Brief Title: "Program "Cerdanya on Fitness" to Improve the Lifestyle of People With Obesity in Cerdanya (CF).
Acronym: CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital of Cerdanya, Spain (Unknown)
Responsible Party: Principal Investigator, Marta Prats Arimon, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2038
Record Dates: First submitted 2022-06-07; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Obesity
Keywords: physical activity,; healthy lifestyle; Mental Health
MeSH Terms: conditions — Obesity; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Model pre-post test in intervention group and pre-post usual follow up in control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Physical Activity: Prescription in physical activity include to perform 1 session a week of exercice led by a sports professional, and 2 sessions of authonomus exercice at 60-80% of participants maximum heart rate.
  Nutritional: Visits and checks every 2 months with a nutritionist with the aim of improving healthy eating habits.
  Positive Mental Health: There are 4 group psycho-emotional sessions based on improving self-esteem, self-control, proactive social attitude and conflict resolution
  Interventions: Behavioral: Cerdanya on Fitness
- Control group (No Intervention): Participants follow the habitual controls in nursing consultation. Recomendations of physical activity and diet.

INTERVENTIONS:
Behavioral: Cerdanya on Fitness — The intervention lasts 9 months. The participants will carry out group activities and will be followed individually by the different interdisciplinary professionals. Goals will be set for each visit. Before and after the training there will be an assessment of physical exercise, nutritional and positive mental health habits.
  Arms: Intervention group

SUMMARY:
To evaluate the effectiveness of an intervention program called "Cerdanya on fitness" based on the prescription of physical activity, healthy nutritional habits and the promotion of positive mental health, adapted to people with obesity to improve their lifestyle and psychoemotional wellbeing

DETAILED DESCRIPTION:
Previous phase:Presentation of the protocol to doctors and nurses of the primary health care center.

Phase 1: After being informed about the study and the possible risks, all patients who give their written informed consent will undergo.

-1) 4 weeks of screening to determine eligibility to enter the study. Referral of patients who meet the inclusion/exclusion criteria to enter the Cerdanya on fitness program by the nursing consultation.

Phase I protocol data collection (physical activity scale, positive mental health scale, Mediterranean diet scale, sociodemographic variables will also be collected week 0) Patients who meet the eligibility requirements will be randomized in a non-blinded fashion. (control group and research group) (5 weeks)

weeks 1-2: Initial assessment of physical fitness and dietary habits in the intervention group (blood test- stress test- anthropometry)

week 3-39: Implementation of the intervention (nutritional, physical activity and psychosocial) to the intervention group. The control group will continue with the usual nursing controls in the primary care center.

40-41 week: Final evaluation of the physical condition and eating habits of the intervention group (blood test, stress test, anthropometry): Final data collection of the control and intervention group (physical activity scale, positive mental health scale, Mediterranean diet scale).

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Body Mass Index 30-40

Exclusion Criteria:

* Serious cognitive impairment
* Serious mental disorder
* Impossibility of performing physical activity for medical diagnosis (IAM < 3 months, hemorrhagic stroke < 3 months, major surgery < 3 months)
* Severe mobility difficulties (people with use of devices such as cane, walker, wheelchair..)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of frecuency and intensity of pysical activity | 9 months
  CLASS AF is a rapid classification scale for physical activity. It is measured based on physical activity at work and physical activity in leisure time, taking into account minutes and frequency. From the formula: 2 x L + Ll x frq 2, the person is classified as sedentary, minimally active, mildly active, moderately active or very active.
Change from baseline mediterrainian diet on 14 points on the scale of adherence to the Mediterranean diet. | 9 months
  The scale of adherence to the Mediterranean diet, is a scale based on 14 items where you ask about 7 groups of foods and portions characteristic of this diet. each item must score with a 1 or 0 depending on the fulfilled or not. The sum of the points if it is less than 9 indicates a bad grip if it is equal to or greater than 9 , a good grip
Change from baseline of positive mental health on 39 points of the Positive Mental Health Scale | 9 months
  The SMP multifactorial scale consists of 39 items that are distributed among 6 factors: Personal Satisfaction, Prosocial Attitude, Self-Control, Autonomy, Problem Solving and Self-Update, and Interpersonal Relationship Skills. The evaluation of each item is done with a scale scale ranging from 1 to 4. Being 1, always or almost always, 2, quite often, 3 often and 4, never or almost never. Finally, a score between 39 and 156 is obtained, the higher the score the more positive mental health.
Change from baseline of the BMI of participants. Weight and height will be combined to report BMI in kg/m^2 | 2 months
  Weigh will be mesured with a analogic weighing machine in Kilograms. Participants are mesured only with underwear clouths. Height will be mesured in m^2.
Change from baseline of watter percentage with a bioimpedance scale | 2 months
  Participants are mesured only with underwear clouths on the bioimpedance scale TANITA BC 602
Change from baseline of fat mass percentage with a bioimpedance scale | 2 months
  Participants are mesured only with underwear clouths on the bioimpedance scale TANITA BC 602
Change from baseline of fat free mass percentage with a bioimpedance scale | 2 months
  Participants are mesured only with underwear clouths on the bioimpedance scale TANITA BC 602
change in the baseline of the caryovascular risk index with the waist-hip measurement | 9 months
  The waist-hip ratio (IC-C) is a specific anthropometric measurement to measure the levels of intra-abdominal fat, it relates the perimeter of the waist to that of the hip (in centimeters) and depending on the result it is estimated if there is a certain cardiovascular risk.
  The WHO establishes normal levels of 0.8 in women and 1 in men; higher values would indicate
Change from baseline of fat percentage and fat Kg on anthropometric measurements | 9 months
  The specific anthropometric measurements for people with obesity according to ISAK are 3 skin folds mesured in mm 3 diameters and 2 perimeters (.Waist circumference 1: at rib height, waist circumference 2: 2 cm above the navel.
  The percentage of fat is determined from specific formula. (F Weltman) Mesured in kg and percentage
Change from baseline of muscle percentage and muscle kg on anthropometric measurements | 9 months
  The specific anthropometric measurements for people with obesity according to ISAK are 3 perimeters (triceps muscles, calf muscles, quadriceps muscles) . The percentage of muscle is determined from specific formulas.( F Lee) mesured in kg and percentage
Change from baseline of bone percentage on anthropometric measurements | 9 months
  The specific anthropometric measurements for people with obesity according to ISAK are 3 diameters. The percentage of bone is determined from specific formulas.(F Rocha) Mesured in kg and percentage
Change from baseline of glucose and cholesterol on blood test | 9 months
  Test levels of HDL, LDL, Triglicerids, Cholesterol Total. Mesured in mg/dL
Change from baseline of glucose and cholesterol on blood test | 9 months
  Test levels of glucose. Mesured in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Marta Prats-Arimon, PHD, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Transfronterer de Cerdanya, Puigcerdà, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD when the periode of collecting data is finished.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from June 2020 until the article will be published
Access Criteria: All team researchers from University of Barcelona and Hospital de Cerdanya can share IPD throught SPSS program by corporative mail.All researchers need a password to access the institution's intranet. In addition, a shared folder will be generated where only researchers have access to share other documents

REFERENCES:
- [Background] Prats-Arimon, M., Barceló-Peiró, O., Ribot-Domènech, I., Heras-Ojea, M., Pérez-Chirinos, C., Vilalta-Serarols, C., Fontecha-Valero, B., Puig-Llobet, M. y Lluch-Canut, M.T. (2020).
- See also: Related Info — http://diposit.ub.edu/dspace/handle/2445/2